CLINICAL TRIAL: NCT03085407
Title: Acute Biliary Pancreatitis - Optimal Time for Cholecystectomy: A Prospective Randomized Study
Brief Title: Acute Biliary Pancreatitis - Optimal Time for Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: South Valley University (Other)
Collaborators: Sohag University (Other)
Responsible Party: Principal Investigator, Mohammed Ahmed Omar, Lecturer of GIT surgery and laparoendoscopy, South Valley University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SVU 148
Record Dates: First submitted 2017-03-19; First posted 2017-03-21 (Actual); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: Acute Biliary Pancreatitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- early cholecystectomy (Active Comparator): Early cholecystectomy was done within 48 after admission
  Interventions: Procedure: early cholecystectomy
- delayed cholecystectomy (Sham Comparator): Delayed cholecystectomy was done after 30 days after randomization.
  Interventions: Procedure: delayed cholecystectomy

INTERVENTIONS:
Procedure: early cholecystectomy — cholecystectomy was done within 48 after admission
  Arms: early cholecystectomy
Procedure: delayed cholecystectomy — cholecystectomy was done after 30 days after randomization
  Arms: delayed cholecystectomy

SUMMARY:
In patients with mild gallstone pancreatitis, early cholecystectomy within 48 hours might reduce the risk of recurrent gallstone-related complications, compared with the more commonly used strategy in our locality of conservative management and delayed cholecystectomy. However, evidence to support early cholecystectomy is poor, and concerns exist about an increased risk of cholecystectomy-related complications with this approach. In this study, we aimed to compare the benefits and harms of early versus delayed cholecystectomy in patients with mild biliary pancreatitis.

DETAILED DESCRIPTION:
Inclusion criteria

1. Patient diagnosed with a first attack of mild biliary pancreatitis
2. Age ≥ 18 years
3. American Society of Anesthesiologists (ASA) grade I, II or III
4. a serum C-reactive protein (CRP) concentration less than 100 mg/L,
5. no need for opioid analgesics,
6. normal oral diet tolerance Exclusion criteria

1. chronic pancreatitis 2. alcohol abuse 3. pregnancy The number of patients needed was calculated. Considering a power of 80% and reliability of 0.05, we found that 53 patients should be present in each group. Eligible patients will be randomly divided into two equal groups (Group 1: early cholecystectomy, Group 2: delayed cholecystectomy) according to a computer-generated random numbers.

Procedure Early cholecystectomy was done within 48 after admission. Delayed cholecystectomy was done after 30 days after randomization. All cholecystectomies were done by, or under the direct supervision of, a surgeon who had undertaken at least 100 cholecystectomies in the past 5 years.

ELIGIBILITY:
Inclusion Criteria:

1. Patient diagnosed with a first attack of mild biliary pancreatitis
2. Age ≥ 18 years
3. American Society of Anesthesiologists (ASA) grade I, II or III
4. a serum C-reactive protein (CRP) concentration less than 100 mg/L,
5. no need for opioid analgesics,
6. normal oral diet tolerance

Exclusion Criteria:

* 1. chronic pancreatitis 2. alcohol abuse 3. pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2014-06-01 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
Gallstone related complications | 6 month of onset of pancreatitis
  recurrent pancreatitis, cholecystitis, cholangitis, obstructive choledocholithiasis needing endoscopic retrograde cholangiopancreatography, or gallstone colic

SECONDARY OUTCOMES:
Difficulty of cholecystectomy | up to 3 hours
  the degree of difficulty of the procedureas assessed by the most experienced surgeon on a 0-10 visual analogue scale
Conversion to open cholecystectomy | up to 2 hours
Operative time | up to 10 hours
  from the begging of the operation to recovery of patient
Cholecystectomy related complications | up to 1 month
additional surgical, endoscopic, or radiological intervention | up to 6 month
Gall stones non related complications | up to 6 month
Length of hospital stay of index admission | from admission to discharge of patient, up to 10 days
Number of readmission | up to 6 month
Total length of hospital stay (including readmission) | up to 6 month
The number of patient-reported colics irrespective of readmission | up to 6 month
Need for intensive care unit admission | up to 6 month
Mortality | up to 6 month
  death from gall stone related complication

IPD SHARING:
Plan to Share IPD: No